CLINICAL TRIAL: NCT01253993
Title: Impaired Decision-making in Adolescents: A Vulnerability Factor for the Development of Substance Use and Abuse.
Brief Title: Impaired Decision-making in Adolescents
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: W. Matthys, UMC Utrecht
Other Study IDs: 05-271; ZonMw 31100001 (Other: ZonMw); NIDA DA 16135 (Other: NIDA)
Record Dates: First submitted 2007-03-02; First posted 2010-12-06 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2010-12

CONDITIONS: Adolescent Psychiatry; Antisocial Personality Disorders; Substance-Related Disorders
Keywords: Disruptive Behavior Disorders, Substance abuse,; Iowa Gambling Task, Decision Making.
MeSH Terms: conditions — Antisocial Personality Disorder; Substance-Related Disorders; Attention Deficit and Disruptive Behavior Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
There is clear evidence that aggressive behavior and disruptive behavior disorders (DBD) in middle childhood are associated with an increased risk for substance abuse in adolescence. However, the exact underlying mechanism of this increased risk is unknown. It is likely that a biopsychological vulnerability in some aggressive children and children with DBD makes them liable to substance use and abuse. The investigators hypothesize that deficient decision making is such a biopsychological factor. In this study the investigators aim to test the latter hypothesis by investigating the decision making ability in a group of adolescents with DBD with and without substance use disorders. Decision-making is assessed with the IOWA Gambling Task (GT). This task mimics real-life situations in the way it factors uncertainty, reward and punishment. The GT is specifically designed to assess impaired decision-making in individuals who are unable to learn from their mistakes and make decisions that repeatedly lead to negative consequences. This characteristic may be common to individuals with externalizing disorders such as DBD, psychopathy, and substance use disorders.

DETAILED DESCRIPTION:
This study consists of two substudies with adolescents in the age of 14-21 years. The first study group consist of adolescents with DBD with (n=30) and without (n=30) substance use disorders. These adolescents are recruited from orthopsychiatric, forensic psychiatric, and judicial institutions.

The second study group consists of a) ex-patients of the Utrecht Coping Power Program (UCPP)who previously participated to a follow-up study, and b) ex-patients who were treated as a child at an outpatient clinic of the UMC Utrecht. These latter groups were taken together and subdivided into a group with (n=30) and without (n=30) substance use problems.

For both studies healthy controls (n=80) are recruited. The investigators will start with healthy controls from earlier studies, and those are extented and will serve as control group for both studies.

ELIGIBILITY:
Inclusion Criteria:

* Having a DISC diagnosis DBD

Exclusion Criteria:

* Having the DISC diagnosis Schizophrenia

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: DBD adolescents were recruited from judicial and forensic institutions. Healthy controls consisted of volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2006-04; Primary Completion 2007-06 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Matthys, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Ernst M, Grant SJ, London ED, Contoreggi CS, Kimes AS, Spurgeon L. Decision making in adolescents with behavior disorders and adults with substance abuse. Am J Psychiatry. 2003 Jan;160(1):33-40. doi: 10.1176/appi.ajp.160.1.33. PMID 12505799